CLINICAL TRIAL: NCT03502252
Title: Experimental Evaluation of Semillas de Apego, a Group-based Program to Foster Maternal Mental Health and Early Childhood Development Among Violence Exposed Communities in Colombia.
Brief Title: Experimental Evaluation of Semillas de Apego
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Los Andes, Columbia (Other)
Collaborators: Genesis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UANDES835
Record Dates: First submitted 2018-04-10; First posted 2018-04-18 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: Child Development; Attachment Disorder; Exposure to Violent Event; Parenting
Keywords: early childhood development; social and emotional development; secure parenting relationships

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Semillas de Apego is a group-based psychosocial program for victimized caregivers with children 2 to 5 in Colombia, a country devastated by violence. The program's builds upon scientific evidence on (i) the way in which violence hinders early childhood development and erodes mothers' mental health and their capacity to form nurturing relationships with their children, and (ii) the effectiveness of promoting healthy child-parent attachments to mitigate the effects of toxic stress on toddlers (Lieberman and Van Horn, 2011).
  Interventions: Behavioral: Semillas de Apego
- Control Group (No Intervention): Centers and participants assigned to the this group continue to have access to the regular early childhood programs offered through the centers to which children are affiliated.

INTERVENTIONS:
Behavioral: Semillas de Apego — Group-based Primary Caregiver Intervention: Group-based psychosocial program for victimized mothers (or alternative primary caregivers) with children 2 to 5, that aims at promoting healthy child-parent attachments as a pathway for a proper development among children exposed to violence.
  Arms: Treatment Group

SUMMARY:
The current trial focuses on the effectiveness evaluation of Semillas de Apego in Tumaco, a municipality in Colombia heavily affected by violence and poverty. Over a time-span of 23 months, the researchers will follow the implementation of Semillas de Apego with 40 groups of 16 participants each, all of them mothers or primary caregivers of children 2 to 5. This will allow the researchers to reach a total of 640 participants and their children. The impact evaluation will be based on a cluster- randomized control trial in which the researchers will assign 1280 eligible subjects, nested within 18 child development centers, to either an intervention arm or a control group. The former group will participate in 15 group-led session over the period of 3 months; the latter will continue to have access to the regular early childhood programs offered through the centers to which children are affiliated. Data will be collected at baseline and two follow-ups: 1 and 12 months after the implementation has concluded. The researchers hypothesize that the program will have a positive and sequential impact on the following dimensions: (i) primary caregiver's mental health, (ii) child rearing practices, (iii) quality of child-parent emotional bond, (iv) children's mental health, and (v) children's cognitive and socioemotional development.

DETAILED DESCRIPTION:
Over half a million children between 0 and 5 years of age in Colombia have been affected by a civil conflict that has spanned over six decades. Exposure to violence during early childhood, or being born to a household that has been formerly victimized, may have devastating consequences on early childhood cognitive and socio-emotional development. In doing so, violence can compromise the right to lead healthy and productive lives for thousands of children in Colombia.

First, violence leaves a legacy of poverty and psychological trauma (Ibañez & Moya, 2010; Moya, 2018). Children who experienced violence during early childhood lag in cognitive, social, and emotional development, while exposure to violence increases the probability of child neglect (Harker, Moya, & Riveros, 2015; Cuartas, Harker, & Moya, 2015). Protecting children from effects of violence, toxic stress, and deficits in family care is therefore one of the key challenges as Colombia transitions into a post-conflict stage and for the construction of a more equal and peaceful society. More generally, identifying cost effective ways to protect children and children from the effects of violence, toxic stress, and deficits in maternal care is a key challenge in contexts of violence and humanitarian crises.

Recent evidence exploring the effect of interventions to promote positive child-development suggest a promising path through the attention to their caregivers (Singla Kumbakumba, & Aboud, 2015; Rahman et al., 2013). Building from this evidence, in this trial the researchers will evaluate the effectiveness of a group-based psychosocial program (Semillas de Apego) for victimized caregivers with children 2 to 5 in Colombia, a country devastated by violence. The program promotes healthy child-parent attachments as a pathway for a proper development among children exposed to violence. By fostering caregivers' mental health and their capacity to become a source of emotional protection, the intervention helps children reach their full potential amid such traumatic circumstances. Delivered in a 15-week curriculum, Semillas de Apego first provides tools so that victimized caregivers can start processing their own trauma. Then, the program focuses on allowing a proper understanding of the child's development trajectories and how they affected by the experience of adversities (such as violence exposure). Finally, the curriculum works towards fostering positive child-rearing practices. Taken together, Semillas de Apego's curriculum aims to foster the healthy child-parent attachments that promote appropriate affect regulation and healthy emotional development in the midst of adverse circumstances.

The current trial focuses on the effectiveness evaluation of Semillas de Apego in Tumaco, a municipality in Colombia heavily affected by violence and poverty. Over a time-span of 23 months, the researchers will follow the implementation of Semillas de Apego with 40 groups of 16 participants each, all of them mothers or primary caregivers of children 2 to 5. This will allow the researchers to reach a total of 640 participants and their children. The impact evaluation will be based on a cluster- randomized control trial in which 1280 eligible subjects, nested within 18 child development centers, will be assigned to either an intervention arm or a control group. The former group will participate in 15 group-led session over the period of 3 months; the latter will continue to have access to the regular early childhood programs offered through the centers to which children are affiliated. Data will be collected at baseline and two follow-ups: 1 and 12 months after the implementation has concluded. The researchers hypothesize that the program will have a positive and sequential impact on the following dimensions: (i) primary caregiver's mental health, (ii) child rearing practices, (iii) quality of child-parent emotional bond, (iv) children's mental health, and (v) children's cognitive and socioemotional development.

ELIGIBILITY:
Inclusion Criteria:

The experimental evaluation of Semillas de Apego will be conducted as a Cluster-Randomized Control Trial (C-RCT). The eligible population for the study are all families served by Genesis Foundation's Early Childhood Development Center (ECDC) in Tumaco, Colombia and whose children's ages range between 2 to 4 years of age. For example, for the first cohort, the children should have been born between August 1st, 2014 to April 1st, 2016

Exclusion Criteria:

None

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1280 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Primary caregiver's mental health | 1 month after the end of intervention
  Measured with four sub-scales of the Symptom Checklist-90-R (Derogatis, 1994).
Child rearing practices | 1 month after the end of intervention
  Measured with a measure asking caregivers whether they engaged in any of the following six stimulating activities with their children in the previous week: (1) reading stories or looking at books with images; (2) telling stories; (3) singing songs; (4) playing with child; (5) taking the child outside; and (6) spending time in physical activities with child. To analyze this construct as a composite measure, the researchers will computed a summary score ranging from zero (no engagement in any activity) to six (engagement in the six activities)
Healthy child-parent emotional bonds | 1 month after the end of intervention
  Measured with the parenting stress-index (PSI, Adibin, 2012), a measure focused on three major domains of stress: child characteristics, parent characteristics and situational/demographic life stress. The researchers will analyze a composite measure of this scale and the individual sub-scales for the following domains: (i) parental distress, (ii) parent-child dysfunctional interaction, and (iii) difficult child.
Children's mental health | 12 months after the end of the intervention
  Measured with two separated scales reported by the caregiver. First, the researchers will employ an adapted measure of the Trauma Symptom Checklist for Young Children (TSCYC, Briere,2005) to describe child-levels of trauma and abuse-related symptomatology. Second, the researchers will employ the brief version of the Infant Toddler Social Emotional Assessment (BITSEA, Carter & Briggs-Gowan, 2004) to screen for social, emotional, and behavioral problems in our population. For both scales, the researchers will focus on composite scores, but also provide detailed findings for each subscale.
Children's cognitive, social, and emotional development | 12 months after the end of the intervention
  Measured with the international Development Learning Assessment (IDELA, Pisani, Borisova & Dowd, 2015). This direct assessment tool, will describe the: (i) motor development, (ii) emergent language and literacy, (iii) emergent numeracy and problem solving, and (iv) socio-emotional skills of children.
Healthy child-parent emotional bonds | 12 months after the end of the intervention
  Measured with an observation measured designed for this trial, this measure will describe the quality of the relationship between children and caregivers in the child-development center. An overall score will be produced and analyzed from observers' ratings to items targeting: (a) the quality of the interaction, (b) the cognitive stimulation provided in the situation, and (c) the emotional support provided during the situation.

SECONDARY OUTCOMES:
Children's mental health: | 1 month after end of the intervention
  Measured with two separated scales reported by the caregiver. First, the researchers will employ an adapted measure of the Trauma Symptom Checklist for Young Children (TSCYC, Briere,2005) to describe child-levels of trauma and abuse-related symptomatology. Second, the researchers will employ the brief version of the Infant Toddler Social Emotional Assessment (BITSEA, Carter & Briggs-Gowan, 2004) to screen for social, emotional, and behavioral problems in our population. For both scales, the researchers will focus on composite scores, but will also provide detailed findings for each subscale.
Children's social, and emotional development. | 1 month after end of the intervention
  Measured at baseline with an adapted version of the Preschool Self-Regulatory Assessment (PSRA, Smith-Donald, Raver, Hayes & Richardson, 2007). This tool will provide independent scores of self-regulations in emotional, attentional, and behavioral domains. The researchers will focus our report on a composite score, but also provide detailed findings for each subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Andres Moya, Ph.D, Principal Investigator — Universidad de Los Andes
Locations (1):
- Semillas de Apego, Tumaco, Departamento de Nariño, Colombia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Data will be available upon publication of the main evaluation article.

DOCUMENTS (1):
  • Study Protocol (2018-03-09): https://cdn.clinicaltrials.gov/large-docs/52/NCT03502252/Prot_000.pdf